CLINICAL TRIAL: NCT05121480
Title: A Phase 2, Multicenter, Double-Blind, Placebo-Controlled, Multiple-Cohort Study Investigating the Effect of EDP1815 in Participants for the Treatment of Mild, Moderate and Severe Atopic Dermatitis
Brief Title: A Study Investigating the Effect of EDP1815 in the Treatment of Mild, Moderate and Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDP1815-207; 2021-001805-63 (EudraCT Number)
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis
Keywords: Mild Atopic Dermatitis; Moderate Atopic Dermatitis; Severe Atopic Dermatitis; Mild Eczema; Moderate Eczema; Severe Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: Cohorts 1, 2 & 3 will be run concurrently, and Cohort 4 recruitment will commence after enrollment for Cohorts 1, 2, & 3 are completed. Randomization to Cohort 4 will not start before randomization to Cohorts 1, 2 & 3 have completed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 100 participants with mild, moderate or severe Atopic Dermatitis 75 participants on EDP1815 and 25 participants on matching placebo administered as 2 capsules (1.6 x 10^11 total cells) once daily for 16 weeks
  Interventions: Drug: EDP1815; Drug: Placebo
- Cohort 2 (Experimental): 100 participants with mild, moderate or severe Atopic Dermatitis 75 participants on EDP1815 and 25 participants on matching placebo administered as 2 capsules (6.4 x 10^11 total cells) once daily for 16 weeks
  Interventions: Drug: EDP1815; Drug: Placebo
- Cohort 3 (Experimental): 100 participants with mild, moderate or severe Atopic Dermatitis 75 participants on EDP1815 and 25 participants on matching placebo administered as 1 capsule (3.2 x 10^11 cells) twice daily (6.4 x 10^11 total cells) for 16 weeks
  Interventions: Drug: EDP1815; Drug: Placebo
- Cohort 4 (Experimental): 105 participants with mild, moderate or severe Atopic Dermatitis 70 participants on EDP1815 and 35 participants on matching placebo administered at 1 capsule (8.0x10^10 total cells) once daily for 16 weeks
  Interventions: Drug: EDP1815; Drug: Placebo

INTERVENTIONS:
Drug: EDP1815 — EDP1815 is an orally administered, pharmaceutical preparation of a single strain of bacteria
  Other Names: Prevotella histicola
Drug: Placebo — Placebo oral capsule

SUMMARY:
The purpose of this research study is to determine whether the study drug, EDP1815, is safe and effective in the treatment of atopic dermatitis compared with placebo. The study will look at different doses of the study drug, and whether there are differences when the drug is given once daily or twice daily.

DETAILED DESCRIPTION:
Atopic dermatitis (atopic eczema) is a very common type of skin disease. It typically causes red, dry, and itchy skin and may have a significant impact on quality of life. Rashes may appear on the arms and behind the knees, or anywhere else on the body. While there are existing therapies, there is currently no cure for atopic dermatitis.

This is a randomized, double blind, placebo controlled, parallel group, Phase 2 study to evaluate the efficacy and safety of EDP1815 in adult participants 18 to ≤75 years of age with mild, moderate, and severe atopic dermatitis (AD).

Participants will be screened within 28 days prior to the first dose of study intervention to confirm study eligibility. Subjects must have mild, moderate, or severe AD involving at least 5% Body Surface Area (BSA); an Investigator Global Assessment (IGA) score of 2, 3, or 4; and an Eczema Area Severity Index (EASI) of at least 6 at screening and Day 1.

All participants must agree to use a background therapy (per protocol) twice daily for at least 14 days prior to Day 1 in order to be considered eligible for the study.

Approximately 405 participants will be randomized to receive either EDP1815 or placebo (295 to EDP1815: 110 to placebo) and treated for 16 weeks. Participants in Cohorts 1, 2, & 3 will be randomized in a 3:1 ratio (225 to EDP1815: 75 to placebo). Participants in Cohort 4 will be randomized in a 2:1 ratio (70 to EDP1815: 35 to placebo). Cohorts 1, 2 & 3 will be run concurrently, and Cohort 4 recruitment will commence after enrollment for Cohorts 1, 2, & 3 are completed.

Randomization will be stratified by baseline disease severity (mild [IGA = 2], moderate [IGA = 3] or severe [IGA = 4] AD). The investigational product will be administered either once or twice daily for 16 weeks. Background emollient (moisturizer) therapy must continue at least twice daily for the duration of the treatment and follow-up periods. Topical rescue therapy is allowed during the treatment period per protocol.

The primary efficacy endpoint is achievement of an EASI-50 response at Week 16. Secondary efficacy endpoints will look at EASI, IGA, BSA, SCORAD, DLQI, Pruritus-NRS, Sleep Disturbance-NRS, POEM, and the need for rescue therapy at Weeks 4, 8, 12 and 16 (unless otherwise specified in the protocol). Safety and efficacy assessments will be conducted at the investigator site by a clinical assessor blinded to treatment assignment. Scheduled clinic study visits for all subjects will occur at Screening, Day 1, Week 2, Week 4, Week 8, Week 12, Week 16 (end of treatment) and Week 20 (post-treatment follow-up). Participants discontinuing early from the study will undergo a 28-day follow-up period, where possible.

At the end of the 16-week study treatment, qualified participants completing the study will have the option to enter an open label study.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Must meet age criteria.
* Must have a diagnosis of atopic dermatitis (AD)for at least 6 months.
* Must have severity of atopic dermatitis meeting the below criteria at both Screening and Day 1:

  * An IGA of 2, 3 or 4 on the vIGA scale, and;
  * A BSA of ≥5%, and;
  * An EASI score of ≥6.
* Must agree to use emollients.
* Must meet contraception requirements.

Exclusion Criteria:

* Have been in a clinical trial for EDP1815 prior to signing of ICF.
* Use of phototherapy or tanning beds; systemic medications/treatments that could affect AD or its symptoms including immunosuppressive therapy (e.g., oral or injectable corticosteroids, methotrexate, azathioprine, cyclosporine, mycophenolate mofetil, JAK inhibitors, tacrolimus, and/or leukotriene inhibitor) within 4 weeks of randomization.
* Treatment with topical agents that could affect atopic dermatitis, including topical corticosteroids, topical calcineurin inhibitors (e.g., tacrolimus or pimecrolimus), or topical PDE-4 inhibitor (e.g., crisaborole) within 14 days prior to randomization.
* Clinically significant abnormalities in screening laboratory values that in the opinion of the Investigator would make a participant unsuitable for inclusion in the study. One retest is permitted within the 28-day screening window.
* Hypersensitivity to P histicola or to any of the excipients.
* Unwillingness to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator.
* Have any other conditions, which, in the opinion of the Investigator or Sponsor, would make the participant unsuitable for inclusion or could interfere with the participant participating in or completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Ehst, MD, PhD, Principal Investigator — Oregon Medical Research Center; Yanislav Mihaylov, MD, Study Director — Evelo Biosciences, Inc.
Locations (59):
- United States (27):
  - USA-131, Birmingham, Alabama
  - USA-112, Fountain Valley, California
  - USA-123, Fremont, California
  - USA-114, Newport Beach, California
  - USA-101, Fort Lauderdale, Florida
  - USA-124, Jacksonville, Florida
  - USA-108, Miami, Florida
  - USA-120, Miami, Florida
  - USA-105, Miramar, Florida
  - USA-102, Orlando, Florida
  - USA-115, Sweetwater, Florida
  - USA-126, Tampa, Florida
  - USA-106, Tampa, Florida
  - USA-118, Sandy Springs, Georgia
  - USA-111, Clarksville, Indiana
  - USA-116, Louisville, Kentucky
  - USA-119, Baton Rouge, Louisiana
  - USA-109, Metairie, Louisiana
  - USA-125, Silver Spring, Maryland
  - USA-130, Ann Arbor, Michigan
  - USA-121, Columbus, Ohio
  - USA-128, Concord, Ohio
  - USA-104, Portland, Oregon
  - USA-127, Memphis, Tennessee
  - USA-117, Frisco, Texas
  - USA-110, Pflugerville, Texas
  - USA-113, Bellevue, Washington
- Australia (4):
  - AUS-102, Carlton
  - AUS-104, Kogarah
  - AUS-101, Melbourne
  - AUS-106, Woolloongabba
- Bulgaria (5):
  - BGR-105, Pleven
  - BGR-104, Sevlievo
  - BGR-101, Sofia
  - BGR-102, Sofia
  - BGR-103, Sofia
- Canada (9):
  - CAN-109, Barrie
  - CAN-108, Edmonton
  - CAN-105, Markham
  - CAN-104, Mississauga
  - CAN-101, Ottawa
  - CAN-107, Richmond Hill
  - CAN-103, Surrey
  - CAN-106, Waterloo
  - CAN-111, Winnipeg
- Germany (7):
  - DEU-105, Berlin
  - DEU-107, Bochum
  - DEU-106, Erlangen
  - DEU-102, Frankfurt am Main
  - DEU-104, Gera
  - DEU-101, Hamburg
  - DEU-103, Heidelberg
- Poland (7):
  - POL-104, Gdansk
  - POL-106, Gdynia
  - POL-107, Katowice
  - POL-105, Lodz
  - POL-101, Lublin
  - POL-102, Warsaw
  - POL-103, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Placebo; Cohort 2 - Placebo; Cohort 3 - Placebo; Cohort 4 - Placebo: Participants with mild, moderate or severe Atopic Dermatitis who received placebo oral capsules.
- Cohort 1 - Active: Participants with mild, moderate or severe Atopic Dermatitis who received 2 capsules (1.6 x 10^11 total cells) of EDP1815 (an orally administered, pharmaceutical preparation of a single strain of bacteria) once daily for 16 weeks.
- Cohort 2 - Active: Participants with mild, moderate or severe Atopic Dermatitis who received 2 capsules (6.4 x 10^11 total cells) of EDP1815 (an orally administered, pharmaceutical preparation of a single strain of bacteria) once daily for 16 weeks.
- Cohort 3 - Active: Participants with mild, moderate or severe Atopic Dermatitis who received 1 capsule (3.2 x 10^11 cells) twice daily (6.4 x 10^11 total cells) of EDP1815 (an orally administered, pharmaceutical preparation of a single strain of bacteria) once daily for 16 weeks.
- Cohort 4 - Active: Participants with mild, moderate or severe Atopic Dermatitis who received 1 capsule (8.0x10^10 total cells) of EDP1815 (an orally administered, pharmaceutical preparation of a single strain of bacteria) once daily for 16 weeks.
Period: Overall Study
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Active | Cohort 2 - Placebo | Cohort 2 - Active | Cohort 3 - Placebo | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Started | 25 | 74 | 25 | 74 | 25 | 86 | 38 | 74
Completed | 19 | 56 | 22 | 53 | 20 | 65 | 36 | 57
Not Completed | 6 | 18 | 3 | 21 | 5 | 21 | 2 | 17
Not completed — Lack of Efficacy | 2 | 2 | 1 | 4 | 0 | 1 | 0 | 2
Not completed — Treatment Failure | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 5 | 3 | 2 | 0 | 4
Not completed — Withdrawal by Subject | 4 | 9 | 1 | 8 | 0 | 9 | 0 | 4
Not completed — Non-compliance with the protocol | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 1
Not completed — Lost to Follow-up | 0 | 4 | 1 | 3 | 1 | 1 | 1 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other Reason | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Active | Cohort 2 - Placebo | Cohort 2 - Active | Cohort 3 - Placebo | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active | Total
Number analyzed (Participants) | 25 | 74 | 25 | 74 | 25 | 86 | 38 | 74 | 421
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (14.79) | 36.1 (16.08) | 42.9 (14.27) | 37.6 (14.38) | 40.2 (17.35) | 39.6 (14.72) | 38.6 (14.78) | 42.7 (14.97) | 39.3 (15.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 36 | 16 | 37 | 10 | 37 | 19 | 43 | 213
  Male | 10 | 38 | 9 | 37 | 15 | 49 | 19 | 31 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 6 | 0 | 2 | 3 | 4 | 22
  Not Hispanic or Latino | 22 | 72 | 23 | 68 | 23 | 84 | 35 | 69 | 396
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 9 | 3 | 9 | 1 | 8 | 4 | 11 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 9 | 4 | 8 | 1 | 7 | 5 | 14 | 51
  White | 19 | 55 | 16 | 55 | 22 | 65 | 26 | 49 | 307
  More than one race | 0 | 1 | 2 | 1 | 0 | 4 | 3 | 0 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 11 | 5 | 16 | 7 | 13 | 12 | 15 | 84
  United States | 8 | 19 | 9 | 20 | 4 | 24 | 10 | 27 | 121
  Poland | 8 | 22 | 6 | 16 | 6 | 23 | 10 | 22 | 113
  Australia | 0 | 2 | 0 | 1 | 1 | 8 | 0 | 2 | 14
  Bulgaria | 3 | 11 | 4 | 12 | 5 | 11 | 3 | 6 | 55
  Germany | 1 | 9 | 1 | 9 | 2 | 7 | 3 | 2 | 34
Baseline IGA Score [Count of Participants; unit: Participants] — The Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA) was use to describe the overall appearance of lesions at a given time-point. The vIGA score ranges from 0 (clear skin) to 4 (severe disease). In order to be eligible for this study, participants had to have a vIGA score of 2, 3, or 4 to participate.
  Participants
    IGA 2 | 4 | 13 | 4 | 12 | 4 | 10 | 7 | 13 | 67
    IGA 3 | 17 | 50 | 17 | 51 | 17 | 64 | 26 | 54 | 296
    IGA 4 | 4 | 11 | 4 | 11 | 4 | 11 | 5 | 7 | 57
Baseline EASI Score [Mean (Standard Deviation); unit: EASI Score] — The Eczema Area Severity Index (EASI) is a validated measure of eczema severity, which considers a combination of the disease severity and body surface area affected across 4 body regions (arms, legs, trunk, and head/neck). The EASI score ranges from 0 - 72, with a lower score indicating a better outcome.
  EASI Score | 15.08 (5.851) | 16.57 (9.420) | 13.74 (5.660) | 16.25 (8.535) | 15.39 (10.175) | 18.07 (10.905) | 15.40 (9.142) | 13.30 (8.049) | 15.81 (9.110)
Baseline BSA [Mean (Standard Deviation); unit: percentage of BSA] — The Body Surface Area (BSA) is a measure of the extent of atopic dermatitis at a given time. It is calculated by estimating the number of participant's handprints of active atopic dermatitis are present where one handprint represents 1% body surface area. This higher the BSA %, the more active atopic dermatitis is present.
  percentage of BSA | 19.78 (12.304) | 23.16 (15.036) | 17.92 (9.939) | 22.76 (15.069) | 21.08 (17.518) | 24.96 (18.291) | 21.86 (18.053) | 19.11 (14.651) | 22.03 (15.780)
Time Since Diagnosis [Mean (Standard Deviation); unit: years] | 20.30 (13.308) | 19.59 (15.221) | 21.82 (18.216) | 18.91 (14.111) | 20.79 (16.586) | 21.44 (16.960) | 24.93 (16.592) | 23.95 (17.248) | 21.34 (16.057)

OUTCOME MEASURES:

1. Primary Outcome: Achievement of EASI-50
Description: The efficacy of EDP1815 will be measured by achieving a decrease of at least 50% from baseline in Eczema Area Severity Index (EASI) score of 50 (EASI-50) at Week 16. The EASI is a validated measure of eczema severity, which considers a combination of the disease severity and body surface area affected across 4 body regions. The EASI score ranges from 0 - 72. A lower score indicates a better outcome.
Time Frame: 16 weeks
Population: Randomized participants who completed the EASI at Week 16 or dropped out before Week 16 for treatment-related reasons.
Measure: Count of Participants; unit: Participants
Groups:
- Cohorts 1-3 - Placebo: Placebo participants from Cohorts 1-3
- Cohort 1 - Active: Mild, moderate or severe Atopic Dermatitis participants taking 2 capsules (1.6 x 10^11 total cells) of EDP1815 once daily for 16 weeks.
- Cohort 2 - Active: Mild, moderate or severe Atopic Dermatitis participants receiving 2 capsules (6.4 x 10^11 total cells) of EDP1815 once daily for 16 weeks.
- Cohort 3 - Active: Mild, moderate or severe Atopic Dermatitis participants receiving 1 capsule (3.2 x 10^11 cells) twice daily (6.4 x 10^11 total cells) of EDP1815 for 16 weeks.
- Cohort 4 - Placebo: Placebo participants from Cohort 4
- Cohort 4 - Active: Mild, moderate or severe Atopic Dermatitis participants receiving 1 capsule (8.0x10^10 total cells) of EDP1815 once daily for 16 weeks.
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 68 | 66 | 66 | 73 | 38 | 66
Participants | 38 | 27 | 25 | 23 | 17 | 25

2. Secondary Outcome: Percentage of Participants Achieving EASI-50
Description: The efficacy of EDP1815 will be measured by the number of participants achieving an EASI-50 at Weeks 4, 8 and 12. The Eczema Area Severity Index (EASI) is a validated measure of eczema severity, which considers a combination of the disease severity and body surface area affected across 4 body regions (arms, legs, trunk, and head/neck). The EASI score ranges from 0 - 72, with a lower score indicating a better outcome.
Time Frame: 4, 8 and 12 weeks
Population: Randomized participants who completed the EASI at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Count of Participants; unit: Participants
Groups:
- Cohorts 1-3 - Placebo: Placebo participants from Cohorts 1, 2 and 3
- Cohort 1 - Active: Mild, moderate or severe Atopic Dermatitis participants received 2 capsules (1.6 x 10^11 total cells) of EDP1815 once daily for 16 weeks.
- Cohort 2 - Active: Mild, moderate or severe Atopic Dermatitis participants received 2 capsules (6.4 x 10^11 total cells) of EDP1815 once daily for 16 weeks.
- Cohort 3 - Active: Mild, moderate or severe Atopic Dermatitis participants on receiving 1 capsule (3.2 x 10^11 cells) twice daily (6.4 x 10^11 total cells) of EDP1815 for 16 weeks.
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 72
Participants
  Week 4: number analyzed (Participants) | 69 | 72 | 70 | 79 | 38 | 70
  Week 4 | 20 | 18 | 14 | 18 | 8 | 23
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 38 | 66
  Week 8 | 23 | 29 | 21 | 22 | 16 | 27
  Week 12: number analyzed (Participants) | 69 | 68 | 66 | 76 | 38 | 64
  Week 12 | 26 | 33 | 21 | 24 | 17 | 24

3. Secondary Outcome: Percentage of Participants Achieving EASI-75
Description: The efficacy of EDP1815 will be measured by the number of participants achieving an EASI-75 at Weeks 4, 8, 12 and 16. The Eczema Area Severity Index (EASI) is a validated measure of eczema severity, which considers a combination of the disease severity and body surface area affected across 4 body regions (arms, legs, trunk, and head/neck). The EASI score ranges from 0 - 72, with a lower score indicating a better outcome.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 72
Participants
  Week 4: number analyzed (Participants) | 69 | 72 | 70 | 79 | 38 | 70
  Week 4 | 1 | 9 | 4 | 6 | 2 | 7
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 38 | 66
  Week 8 | 5 | 11 | 11 | 9 | 9 | 11
  Week 12: number analyzed (Participants) | 69 | 68 | 66 | 76 | 38 | 64
  Week 12 | 11 | 13 | 8 | 13 | 10 | 15
  Week 16: number analyzed (Participants) | 68 | 66 | 66 | 73 | 38 | 66
  Week 16 | 22 | 13 | 9 | 13 | 9 | 11

4. Secondary Outcome: Percentage of Participants Achieving EASI-90
Description: The efficacy of EDP1815 will be measured by the number of participants achieving an EASI-90 at Weeks 4, 8, 12 and 16. The Eczema Area Severity Index (EASI) is a validated measure of eczema severity, which considers a combination of the disease severity and body surface area affected across 4 body regions (arms, legs, trunk, and head/neck). The EASI score ranges from 0 - 72, with a lower score indicating a better outcome.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 72
Participants
  Week 4: number analyzed (Participants) | 69 | 72 | 70 | 79 | 38 | 70
  Week 4 | 0 | 3 | 1 | 1 | 0 | 1
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 38 | 66
  Week 8 | 1 | 3 | 3 | 4 | 2 | 4
  Week 12: number analyzed (Participants) | 69 | 68 | 66 | 76 | 38 | 64
  Week 12 | 6 | 5 | 5 | 3 | 4 | 7
  Week 16: number analyzed (Participants) | 68 | 66 | 66 | 73 | 38 | 66
  Week 16 | 8 | 3 | 5 | 6 | 1 | 4

5. Secondary Outcome: Mean Absolute Change in EASI
Description: The efficacy of EDP1815 will be measured using the mean absolute change from baseline in EASI at weeks 4, 8, 12 and 16. The Eczema Area Severity Index (EASI) is a validated measure of eczema severity, which considers a combination of the disease severity and body surface area affected across 4 body regions (arms, legs, trunk, and head/neck). The EASI score ranges from 0 - 72, with a lower score indicating a better outcome.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 71 | 76 | 38 | 69
score on a scale
  Week 4: number analyzed (Participants) | 68 | 69 | 67 | 73 | 34 | 65
  Week 4 | -2.88 (5.229) | -4.57 (6.248) | -1.87 (7.020) | -3.72 (7.947) | -3.09 (5.834) | -3.36 (5.293)
  Week 8: number analyzed (Participants) | 69 | 68 | 67 | 72 | 36 | 62
  Week 8 | -4.30 (5.642) | -5.68 (6.823) | -3.05 (8.001) | -4.54 (8.930) | -5.57 (6.665) | -4.22 (5.056)
  Week 12: number analyzed (Participants) | 69 | 68 | 64 | 71 | 37 | 60
  Week 12 | -5.42 (5.590) | -6.38 (7.924) | -3.56 (8.049) | -5.12 (8.982) | -6.58 (6.758) | -4.82 (5.063)
  Week 16: number analyzed (Participants) | 68 | 66 | 64 | 69 | 38 | 63
  Week 16 | -6.48 (6.360) | -5.83 (7.915) | -4.55 (7.897) | -5.11 (9.116) | -6.99 (6.806) | -4.82 (5.480)

6. Secondary Outcome: Mean Percentage Change in EASI
Description: The efficacy of EDP1815 will be measured using the mean percentage change from baseline in EASI from baseline at weeks 4, 8, 12 and 16. The Eczema Area Severity Index (EASI) is a validated measure of eczema severity, which considers a combination of the disease severity and body surface area affected across 4 body regions (arms, legs, trunk, and head/neck). The EASI score ranges from 0 - 72, with a lower score indicating a better outcome.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 71 | 76 | 38 | 69
percentage change from baseline
  Week 4: number analyzed (Participants) | 68 | 69 | 67 | 73 | 34 | 65
  Week 4 | -20.13 (36.926) | -27.36 (38.993) | -13.96 (48.008) | -22.80 (40.131) | -23.30 (35.369) | -27.30 (41.493)
  Week 8: number analyzed (Participants) | 69 | 68 | 67 | 72 | 36 | 62
  Week 8 | -30.96 (36.521) | -35.33 (42.920) | -22.70 (50.991) | -27.14 (43.544) | -43.08 (36.432) | -35.92 (40.244)
  Week 12: number analyzed (Participants) | 69 | 68 | 64 | 71 | 37 | 60
  Week 12 | -40.05 (38.450) | -38.40 (48.605) | -24.69 (49.969) | -31.95 (44.916) | -44.99 (34.922) | -41.28 (40.377)
  Week 16: number analyzed (Participants) | 68 | 66 | 64 | 69 | 38 | 63
  Week 16 | -46.97 (44.193) | -35.72 (49.737) | -31.03 (46.957) | -32.68 (45.752) | -45.58 (35.526) | -39.35 (39.316)

7. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (vIGA) of 0 or 1 With a ≥2 Point Improvement
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a vIGA of 0 or 1 with a ≥2 Point Improvement from baseline at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: Randomized participants who completed the vIGA at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 72
Participants
  Week 4: number analyzed (Participants) | 69 | 72 | 70 | 79 | 38 | 70
  Week 4 | 1 | 5 | 3 | 2 | 2 | 4
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 38 | 66
  Week 8 | 3 | 5 | 5 | 6 | 5 | 9
  Week 12: number analyzed (Participants) | 69 | 68 | 66 | 76 | 38 | 64
  Week 12 | 6 | 6 | 5 | 6 | 6 | 9
  Week 16: number analyzed (Participants) | 68 | 65 | 66 | 74 | 38 | 66
  Week 16 | 12 | 5 | 7 | 10 | 2 | 7

8. Secondary Outcome: Percentage of Participants Achieving vIGA of 0 or 1
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a vIGA of 0 or 1 at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 72
Participants
  Week 4: number analyzed (Participants) | 69 | 72 | 70 | 79 | 38 | 70
  Week 4 | 2 | 7 | 3 | 4 | 3 | 8
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 38 | 66
  Week 8 | 4 | 7 | 5 | 7 | 8 | 12
  Week 12: number analyzed (Participants) | 69 | 68 | 66 | 76 | 38 | 64
  Week 12 | 12 | 10 | 5 | 9 | 9 | 11
  Week 16: number analyzed (Participants) | 68 | 65 | 66 | 74 | 38 | 66
  Week 16 | 19 | 10 | 7 | 11 | 5 | 9

9. Secondary Outcome: Percentage of Participants Achieving vIGA of 0
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a vIGA of 0 at Week16
Time Frame: 16 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 68 | 65 | 66 | 74 | 38 | 66
Participants | 2 | 1 | 2 | 1 | 0 | 3

10. Secondary Outcome: Mean Absolute Change in vIGA*BSA
Description: The efficacy of EDP1815 will be measured using the mean absolute change from baseline in vIGA (Validated Investigator Global Assessment) multiplied by the BSA (body surface area) at weeks 4, 8, 12 and 16.
Time Frame: 4, 8, 12, and 16 weeks
Population: Randomized participants who completed the vIGA and BSA at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 71 | 76 | 38 | 69
score on a scale
  Week 4: number analyzed (Participants) | 68 | 69 | 67 | 73 | 34 | 65
  Week 4 | -6.47 (27.832) | -15.84 (33.960) | -5.96 (40.678) | -10.92 (52.802) | -11.04 (29.770) | -14.07 (30.797)
  Week 8: number analyzed (Participants) | 69 | 68 | 67 | 72 | 36 | 62
  Week 8 | -14.49 (36.336) | -21.31 (41.564) | -12.46 (45.651) | -14.53 (59.754) | -21.63 (32.517) | -17.88 (29.523)
  Week 12: number analyzed (Participants) | 69 | 68 | 64 | 71 | 37 | 60
  Week 12 | -20.83 (36.619) | -24.85 (58.901) | -10.48 (45.919) | -17.26 (60.858) | -28.91 (40.904) | -19.56 (30.250)
  Week 16: number analyzed (Participants) | 68 | 65 | 64 | 69 | 38 | 63
  Week 16 | -25.70 (36.633) | -18.90 (58.271) | -14.52 (46.948) | -18.10 (59.953) | -31.00 (42.250) | -24.23 (35.523)

11. Secondary Outcome: Mean Percentage Change in vIGA*BSA
Description: The efficacy of EDP1815 will be measured using the mean percentage change from baseline in vIGA (Validated Investigator Global Assessment) multiplied by the BSA (body surface area) at weeks 4, 8, 12 and 16.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 71 | 76 | 38 | 69
percentage of change
  Week 4: number analyzed (Participants) | 68 | 69 | 67 | 73 | 34 | 65
  Week 4 | -14.82 (47.171) | -21.83 (47.440) | -9.70 (59.410) | -13.26 (75.742) | -19.01 (49.996) | -25.99 (51.487)
  Week 8: number analyzed (Participants) | 69 | 68 | 67 | 72 | 36 | 62
  Week 8 | -25.95 (51.703) | -32.16 (54.509) | -21.27 (65.335) | -15.77 (78.290) | -42.98 (44.572) | -35.85 (47.881)
  Week 12: number analyzed (Participants) | 69 | 68 | 64 | 71 | 37 | 60
  Week 12 | -39.10 (50.435) | -33.23 (74.662) | -18.83 (68.537) | -23.49 (79.946) | -43.64 (52.832) | -37.27 (51.582)
  Week 16: number analyzed (Participants) | 68 | 65 | 64 | 69 | 38 | 63
  Week 16 | -49.25 (51.883) | -28.17 (78.637) | -23.15 (71.749) | -23.74 (81.817) | -44.29 (60.140) | -43.02 (41.198)

12. Secondary Outcome: Mean Absolute Change From Baseline in BSA
Description: The efficacy of EDP1815 will be measured using the mean absolute change from baseline in BSA (body surface area) at weeks 4, 8, 12 and 16. The Body Surface Area (BSA) is a measure of the extent of atopic dermatitis at a given time. It is calculated by estimating the number of participant's handprints of active atopic dermatitis are present where one handprint represents 1% body surface area. This higher the BSA %, the more active atopic dermatitis is present.
Time Frame: 4, 8, 12, and 16 weeks
Population: Randomized participants who completed the BSA at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 71 | 76 | 38 | 69
percentage of BSA
  Week 4: number analyzed (Participants) | 68 | 69 | 67 | 73 | 34 | 65
  Week 4 | -2.06 (7.127) | -3.87 (8.429) | -1.81 (10.573) | -3.09 (13.025) | -2.50 (7.886) | -3.43 (7.503)
  Week 8: number analyzed (Participants) | 69 | 68 | 67 | 72 | 36 | 62
  Week 8 | -3.96 (8.354) | -5.58 (10.766) | -4.10 (12.211) | -4.09 (14.854) | -5.42 (8.712) | -4.50 (8.021)
  Week 12: number analyzed (Participants) | 69 | 68 | 64 | 71 | 37 | 60
  Week 12 | -5.61 (9.432) | -6.79 (14.420) | -3.21 (12.990) | -5.13 (15.342) | -7.96 (11.601) | -5.36 (8.550)
  Week 16: number analyzed (Participants) | 68 | 66 | 64 | 69 | 38 | 63
  Week 16 | -7.18 (9.772) | -5.65 (14.554) | -4.30 (12.902) | -4.96 (15.289) | -8.87 (11.221) | -6.28 (9.078)

13. Secondary Outcome: Mean Percentage Change From Baseline in BSA
Description: The efficacy of EDP1815 will be measured using the mean percentage change from baseline in BSA (body surface area) at weeks 4, 8, 12 and 16. The Body Surface Area (BSA) is a measure of the extent of atopic dermatitis at a given time. It is calculated by estimating the number of participant's handprints of active atopic dermatitis are present where one handprint represents 1% body surface area. This higher the BSA %, the more active atopic dermatitis is present.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 71 | 76 | 38 | 69
percentage change from baseline
  Week 4: number analyzed (Participants) | 68 | 69 | 67 | 73 | 34 | 65
  Week 4 | -12.70 (38.657) | -18.45 (36.769) | -7.55 (48.616) | -12.51 (56.294) | -15.29 (44.347) | -20.56 (36.664)
  Week 8: number analyzed (Participants) | 69 | 68 | 67 | 72 | 36 | 62
  Week 8 | -23.23 (37.106) | -27.19 (44.087) | -20.92 (53.115) | -14.54 (61.187) | -34.23 (41.835) | -28.75 (40.087)
  Week 12: number analyzed (Participants) | 69 | 68 | 64 | 71 | 37 | 60
  Week 12 | -31.79 (45.657) | -30.78 (57.815) | -16.34 (59.085) | -22.17 (61.255) | -39.35 (46.518) | -31.91 (44.645)
  Week 16: number analyzed (Participants) | 68 | 66 | 64 | 69 | 38 | 63
  Week 16 | -41.54 (48.345) | -26.73 (60.521) | -21.74 (56.381) | -20.93 (63.590) | -40.61 (52.352) | -34.81 (37.995)

14. Secondary Outcome: Percentage of Participants Achieving BSA-50
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a BSA-50 at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 72
Participants
  Week 4: number analyzed (Participants) | 69 | 72 | 70 | 79 | 38 | 70
  Week 4 | 12 | 12 | 12 | 17 | 6 | 16
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 38 | 66
  Week 8 | 19 | 21 | 21 | 18 | 15 | 19
  Week 12: number analyzed (Participants) | 69 | 68 | 66 | 76 | 38 | 64
  Week 12 | 23 | 27 | 18 | 20 | 17 | 24
  Week 16: number analyzed (Participants) | 68 | 66 | 66 | 73 | 38 | 66
  Week 16 | 32 | 23 | 19 | 18 | 16 | 20

15. Secondary Outcome: Percentage of Participants Achieving BSA-75
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a BSA-75 at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 72
Participants
  Week 4: number analyzed (Participants) | 69 | 72 | 70 | 79 | 38 | 70
  Week 4 | 4 | 7 | 2 | 2 | 2 | 4
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 38 | 66
  Week 8 | 3 | 11 | 6 | 6 | 6 | 11
  Week 12: number analyzed (Participants) | 69 | 68 | 66 | 76 | 38 | 64
  Week 12 | 11 | 15 | 6 | 10 | 10 | 13
  Week 16: number analyzed (Participants) | 68 | 66 | 66 | 73 | 38 | 66
  Week 16 | 21 | 12 | 8 | 13 | 7 | 12

16. Secondary Outcome: Percentage of Participants Achieving BSA Reduction to 3% BSA or Less
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a BSA reduction to 3% BSA or less at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 72
Participants
  Week 4: number analyzed (Participants) | 69 | 72 | 70 | 79 | 38 | 70
  Week 4 | 3 | 5 | 3 | 4 | 3 | 8
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 38 | 66
  Week 8 | 2 | 8 | 7 | 6 | 10 | 12
  Week 12: number analyzed (Participants) | 69 | 68 | 66 | 76 | 38 | 64
  Week 12 | 12 | 11 | 5 | 8 | 8 | 14
  Week 16: number analyzed (Participants) | 68 | 66 | 66 | 73 | 38 | 66
  Week 16 | 20 | 12 | 7 | 10 | 8 | 10

17. Secondary Outcome: Mean Absolute Change From Baseline in SCORing Atopic Dermatitis (SCORAD)
Description: The efficacy of EDP1815 will be measured using the mean absolute change from baseline in SCORing Atopic Dermatitis (SCORAD) at weeks 4, 8, 12 and 16. The SCORAD is a clinical tool to assess the extent and severity of eczema, to assess treatment effects. There is both an investigator-rated area score using rule of nines to assess disease extent and a disease intensity score comprising erythema, swelling, oozing/crusting, exoriation, lichenification and dryness and a subjective symptoms component which considers itch and sleeplessness scored using a visual analog scale. These scores combine to give a SCORAD score between 0 - 103, with a higher score indicating worse atopic dermatitis.
Time Frame: 4, 8, 12, and 16 weeks
Population: Randomized participants who completed the SCORAD at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cohort 1-3 - Placebo: Placebo participants from Cohorts 1, 2 and 3
Arm/Group | Cohort 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 71 | 71 | 76 | 38 | 71
score on a scale
  Week 4: number analyzed (Participants) | 67 | 67 | 66 | 73 | 33 | 64
  Week 4 | -7.53 (10.655) | -9.79 (14.561) | -5.03 (12.977) | -5.61 (12.761) | -9.57 (13.608) | -8.08 (13.525)
  Week 8: number analyzed (Participants) | 69 | 66 | 67 | 72 | 35 | 60
  Week 8 | -10.92 (13.228) | -11.82 (14.587) | -9.22 (15.082) | -7.45 (16.543) | -14.95 (15.082) | -9.22 (13.271)
  Week 12: number analyzed (Participants) | 69 | 66 | 63 | 71 | 36 | 58
  Week 12 | -15.74 (15.335) | -12.43 (16.200) | -9.19 (15.339) | -9.81 (15.782) | -13.61 (15.179) | -11.16 (14.688)
  Week 16: number analyzed (Participants) | 68 | 64 | 62 | 69 | 38 | 62
  Week 16 | -18.47 (15.920) | -12.05 (16.072) | -11.80 (16.573) | -11.04 (18.009) | -14.58 (16.659) | -11.60 (15.521)

18. Secondary Outcome: Mean Percentage Change From Baseline in SCORAD
Description: The efficacy of EDP1815 will be measured using the mean percentage change from baseline in SCORAD at weeks 4, 8, 12 and 16. The SCORAD is a clinical tool to assess the extent and severity of eczema, to assess treatment effects. There is both an investigator-rated area score using rule of nines to assess disease extent and a disease intensity score comprising erythema, swelling, oozing/crusting, exoriation, lichenification and dryness and a subjective symptoms component which considers itch and sleeplessness scored using a visual analog scale. These scores combine to give a SCORAD score between 0 - 103, with a higher score indicating worse atopic dermatitis.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 71 | 71 | 76 | 38 | 71
percentage change from baseline
  Week 4: number analyzed (Participants) | 67 | 67 | 66 | 73 | 33 | 64
  Week 4 | -15.27 (20.788) | -17.42 (28.161) | -9.30 (27.186) | -11.94 (25.258) | -18.01 (25.219) | -16.43 (26.070)
  Week 8: number analyzed (Participants) | 69 | 66 | 67 | 72 | 35 | 60
  Week 8 | -21.29 (24.598) | -21.74 (29.649) | -17.75 (30.305) | -14.62 (32.958) | -30.08 (29.043) | -20.06 (27.947)
  Week 12: number analyzed (Participants) | 69 | 66 | 63 | 71 | 36 | 58
  Week 12 | -30.92 (28.283) | -22.70 (32.777) | -17.69 (30.135) | -19.71 (31.608) | -27.25 (30.640) | -24.52 (32.251)
  Week 16: number analyzed (Participants) | 68 | 64 | 62 | 69 | 38 | 62
  Week 16 | -36.37 (29.640) | -21.52 (33.038) | -20.96 (31.086) | -20.42 (33.785) | -27.57 (32.326) | -24.10 (32.563)

19. Secondary Outcome: Percentage of Participants Achieving SCORAD-50
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a SCORAD-50 at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 71
Participants
  Week 4: number analyzed (Participants) | 69 | 71 | 69 | 79 | 37 | 69
  Week 4 | 2 | 10 | 4 | 6 | 4 | 8
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 37 | 64
  Week 8 | 6 | 12 | 10 | 9 | 10 | 8
  Week 12: number analyzed (Participants) | 69 | 68 | 65 | 76 | 37 | 62
  Week 12 | 15 | 12 | 7 | 12 | 9 | 11
  Week 16: number analyzed (Participants) | 68 | 66 | 64 | 73 | 38 | 65
  Week 16 | 21 | 8 | 9 | 16 | 10 | 12

20. Secondary Outcome: Percentage of Participants Achieving SCORAD-75
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a SCORAD-75 at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 72 | 73 | 73 | 81 | 38 | 71
Participants
  Week 4: number analyzed (Participants) | 69 | 71 | 68 | 79 | 37 | 69
  Week 4 | 0 | 1 | 0 | 2 | 0 | 1
  Week 8: number analyzed (Participants) | 69 | 69 | 69 | 78 | 37 | 64
  Week 8 | 1 | 2 | 0 | 5 | 3 | 1
  Week 12: number analyzed (Participants) | 69 | 68 | 65 | 76 | 37 | 62
  Week 12 | 5 | 2 | 1 | 2 | 1 | 4
  Week 16: number analyzed (Participants) | 68 | 66 | 64 | 73 | 38 | 65
  Week 16 | 7 | 1 | 1 | 5 | 2 | 4

21. Secondary Outcome: Mean Absolute Change From Baseline in the Dermatology Quality of Life Index (DLQI)
Description: The efficacy of EDP1815 will be measured using the mean absolute change from baseline in the Dermatology Quality of Life Index (DLQI) at weeks 4, 8, 12 and 16. The DLQI is a validated patient reported outcomes instrument comprised of 10 questions to assess how a participant's skin disease has affected their quality of life over the past week. The score ranges from 0 - 30, with a higher score indicating greater impairment of quality of life. A 4-point change from baseline is considered the minimal clinically important difference threshold.
Time Frame: 4, 8, 12, and 16 weeks
Population: Randomized participants who completed the DLQI at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 71 | 72 | 71 | 77 | 38 | 68
score on a scale
  Week 4: number analyzed (Participants) | 66 | 68 | 65 | 73 | 33 | 65
  Week 4 | -2.6 (4.34) | -2.7 (4.93) | -2.4 (4.20) | -2.4 (5.61) | -3.0 (5.77) | -3.1 (6.03)
  Week 8: number analyzed (Participants) | 68 | 67 | 67 | 72 | 36 | 61
  Week 8 | -3.6 (5.27) | -3.4 (6.40) | -3.1 (5.09) | -3.0 (6.39) | -5.1 (6.76) | -3.3 (6.55)
  Week 12: number analyzed (Participants) | 68 | 67 | 63 | 71 | 37 | 58
  Week 12 | -4.2 (5.15) | -3.5 (5.75) | -2.1 (4.78) | -3.7 (5.74) | -4.2 (6.81) | -3.5 (6.95)
  Week 16: number analyzed (Participants) | 67 | 66 | 64 | 70 | 38 | 63
  Week 16 | -5.4 (5.49) | -3.6 (6.47) | -3.5 (5.12) | -3.7 (6.49) | -4.3 (5.78) | -4.5 (6.76)

22. Secondary Outcome: Mean Percentage Change From Baseline in DLQI
Description: The efficacy of EDP1815 will be measured using the mean percentage change from baseline in the DLQI at weeks 4, 8, 12 and 16. The DLQI is a validated patient reported outcomes instrument comprised of 10 questions to assess how a participant's skin disease has affected their quality of life over the past week. The score ranges from 0 - 30, with a higher score indicating greater impairment of quality of life.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 71 | 72 | 71 | 77 | 37 | 68
percentage change from baseline
  Week 4: number analyzed (Participants) | 66 | 68 | 65 | 73 | 32 | 65
  Week 4 | -20.56 (42.424) | -21.97 (43.095) | -19.48 (47.134) | -14.35 (76.350) | -22.67 (52.475) | -10.28 (73.896)
  Week 8: number analyzed (Participants) | 68 | 67 | 67 | 72 | 35 | 61
  Week 8 | -28.63 (57.232) | -27.49 (46.333) | -25.84 (46.946) | -18.56 (84.619) | -30.29 (61.213) | -12.05 (79.431)
  Week 12: number analyzed (Participants) | 68 | 67 | 63 | 71 | 36 | 58
  Week 12 | -31.11 (63.580) | -25.89 (47.527) | -12.86 (65.083) | -27.61 (76.072) | -25.25 (76.866) | -10.44 (84.857)
  Week 16: number analyzed (Participants) | 67 | 66 | 64 | 70 | 37 | 63
  Week 16 | -45.78 (52.438) | -20.13 (67.256) | -29.67 (46.996) | -26.63 (79.367) | -37.04 (49.074) | -17.68 (82.217)

23. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥4 in the DLQI, of Those With a Score of ≥4 at Baseline
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a reduction of ≥4 in the DLQI, of those with a score of ≥4 at baseline at Week 16. The DLQI score ranges from 0 to 30, with higher scores indicating greater impairment of quality of life.
Time Frame: 16 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 61 | 59 | 61 | 71 | 34 | 63
Participants | 40 | 24 | 23 | 30 | 17 | 24

24. Secondary Outcome: Mean Absolute Change From Baseline in Worst Pruritus Numerical Rating Scale (PR-NRS)
Description: The efficacy of EDP1815 will be measured using the mean absolute change from baseline in the worst Pruritus Numerical Rating Scale (PR-NRS) at weeks 4, 8, 12 and 16. The PP-NRS is a scale from 0 ("no itch") to 10 ("worse imaginable itch") for participants to rate their worst itch that they have experienced over the previous 24 hours. The value calculated for each visit is the mean of the daily values for the 7 days on and before the visit date as long as at least 4 non-missing scores are available.
Time Frame: 4, 8, 12, and 16 weeks
Population: Randomized participants who completed the PP-NRS at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 71 | 70 | 68 | 72 | 36 | 63
score on a scale
  Week 4: number analyzed (Participants) | 65 | 65 | 63 | 69 | 29 | 58
  Week 4 | -0.53 (1.933) | -0.45 (1.962) | -0.65 (2.052) | -0.57 (1.692) | -1.52 (1.845) | -0.72 (1.828)
  Week 8: number analyzed (Participants) | 67 | 64 | 64 | 69 | 26 | 52
  Week 8 | -1.18 (2.452) | -1.04 (2.483) | -0.83 (2.103) | -1.17 (1.986) | -1.97 (1.978) | -0.84 (1.856)
  Week 12: number analyzed (Participants) | 64 | 63 | 61 | 67 | 30 | 52
  Week 12 | -1.54 (2.581) | -1.24 (2.613) | -0.99 (2.171) | -1.34 (1.921) | -1.73 (1.955) | -0.95 (2.095)
  Week 16: number analyzed (Participants) | 60 | 59 | 54 | 62 | 28 | 52
  Week 16 | -1.84 (2.454) | -1.35 (2.674) | -1.00 (2.167) | -1.37 (2.218) | -1.91 (2.007) | -1.08 (2.305)

25. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥2 in the Worst Pruritus-NRS, of Those With a Score of ≥2 at Baseline
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a reduction of ≥2 in the worst PR-NRS score, of those with a score of ≥2 at baseline at Weeks 4, 8, 12 and 16. The PP-NRS is a scale from 0 ("no itch") to 10 ("worse imaginable itch") for participants to rate their worst itch that they have experienced over the previous 24 hours.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 70 | 71 | 70 | 78 | 38 | 67
Participants
  Week 4: number analyzed (Participants) | 65 | 68 | 65 | 75 | 35 | 63
  Week 4 | 11 | 14 | 12 | 11 | 10 | 10
  Week 8: number analyzed (Participants) | 66 | 65 | 66 | 75 | 29 | 56
  Week 8 | 21 | 20 | 14 | 20 | 11 | 13
  Week 12: number analyzed (Participants) | 63 | 63 | 63 | 72 | 31 | 57
  Week 12 | 25 | 20 | 15 | 25 | 10 | 13
  Week 16: number analyzed (Participants) | 59 | 61 | 56 | 67 | 29 | 56
  Week 16 | 29 | 18 | 14 | 22 | 12 | 13

26. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥4 in the Worst PR-NRS, of Those With a Score of ≥4 at Baseline
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a reduction of ≥4 in the worst PR-NRS score, of those with a score of ≥4 at baseline at Week 16. The PP-NRS is a scale from 0 ("no itch") to 10 ("worse imaginable itch") for participants to rate their worst itch that they have experienced over the previous 24 hours.
Time Frame: 16 weeks
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 50 | 53 | 50 | 61 | 25 | 47
Participants | 13 | 9 | 5 | 7 | 5 | 3

27. Secondary Outcome: Mean Absolute Change From Baseline in the Sleep Disturbance Numerical Rating Scale (SD-NRS) Score
Description: The efficacy of EDP1815 will be measured using the mean absolute change from baseline in Sleep Disturbance Numerical Rating Scale (SD-NRS) score at weeks 4, 8, 12 and 16. The SD-NRS is a scale from 0 ("best possible sleep") to 10 ("worse possible sleep") for participants to rate their worst sleep that they have experienced over the previous 24 hours. The value calculated for each visit is the mean of the daily values for the 7 days on and before the visit date as long as at least 4 non-missing scores are available.
Time Frame: 4, 8, 12, and 16 weeks
Population: Randomized participants who completed the SD-NRS at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 71 | 70 | 68 | 72 | 36 | 63
score on a scale
  Week 4: number analyzed (Participants) | 65 | 65 | 63 | 69 | 29 | 58
  Week 4 | -0.36 (1.834) | -0.52 (1.872) | -0.27 (1.985) | -0.16 (1.457) | -0.93 (2.226) | -0.11 (2.126)
  Week 8: number analyzed (Participants) | 67 | 64 | 64 | 69 | 26 | 52
  Week 8 | -1.09 (2.342) | -0.97 (2.128) | -0.56 (1.985) | -0.49 (1.840) | -1.28 (1.956) | -0.35 (2.145)
  Week 12: number analyzed (Participants) | 64 | 63 | 61 | 67 | 30 | 52
  Week 12 | -1.24 (2.568) | -1.06 (2.315) | -0.62 (2.003) | -0.58 (1.916) | -1.22 (2.060) | -0.42 (2.369)
  Week 16: number analyzed (Participants) | 60 | 59 | 54 | 62 | 28 | 52
  Week 16 | 01.48 (2.457) | -1.23 (2.336) | -0.77 (1.936) | -0.63 (1.988) | -1.36 (2.102) | -0.51 (2.374)

28. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥2 in SD-NRS Score, of Those With a Score of ≥2 at Baseline
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a reduction of ≥2 in the SD-NRS score, of those with a score of ≥2 at baseline at Week 16. The SD-NRS is a scale from 0 ("best possible sleep") to 10 ("worse possible sleep") for participants to rate their worst sleep that they have experienced over the previous 24 hours.
Time Frame: 16 weeks
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 56 | 54 | 54 | 63 | 25 | 52
Participants | 25 | 16 | 11 | 13 | 8 | 9

29. Secondary Outcome: Mean Absolute Change From Baseline in Patient Oriented Eczema Measure (POEM)
Description: The efficacy of EDP1815 will be measured using the mean absolute change from baseline in the Patient Oriented Eczema Measure (POEM) at weeks 4, 8, 12 and 16. There are 7 questions scored from 0 (no days) to 4 (every day), giving a POEM score range from 0 to 28, with higher scores representing higher disease severity.
Time Frame: 4, 8, 12, and 16 weeks
Population: Randomized participants who completed the POEM at the relevant visit or dropped out before the relevant visit for treatment-related reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 71 | 71 | 71 | 76 | 37 | 68
score on a scale
  Week 4: number analyzed (Participants) | 66 | 67 | 65 | 72 | 33 | 65
  Week 4 | -2.1 (5.48) | -2.4 (5.75) | -1.6 (5.24) | -3.0 (5.57) | -3.1 (5.66) | -2.7 (6.37)
  Week 8: number analyzed (Participants) | 68 | 66 | 67 | 71 | 35 | 62
  Week 8 | -3.7 (6.31) | -3.8 (6.99) | -2.9 (5.80) | -3.3 (5.88) | -5.4 (6.94) | -3.2 (6.80)
  Week 12: number analyzed (Participants) | 68 | 66 | 63 | 70 | 36 | 58
  Week 12 | -5.1 (7.30) | -4.1 (7.58) | -2.0 (5.44) | -3.9 (6.24) | -4.9 (8.38) | -3.5 (7.17)
  Week 16: number analyzed (Participants) | 67 | 65 | 64 | 68 | 37 | 63
  Week 16 | -6.3 (7.20) | -3.7 (7.93) | -3.8 (6.41) | -3.8 (7.32) | -5.5 (7.53) | -4.3 (7.58)

30. Secondary Outcome: Mean Percentage Change From Baseline in Patient Oriented Eczema Measure (POEM)
Description: The efficacy of EDP1815 will be measured using the percentage change from baseline in the Patient Oriented Eczema Measure (POEM) at weeks 4, 8, 12 and 16. There are 7 questions scored from 0 (no days) to 4 (every day), giving a POEM score range from 0 to 28, with higher scores representing higher disease severity.
Time Frame: 4, 8, 12, and 16 weeks
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 75 | 74 | 74 | 86 | 38 | 74
percentage change from baseline
  Week 4: number analyzed (Participants) | 65 | 67 | 66 | 72 | 33 | 65
  Week 4 | -10.43 (35.777) | -12.19 (36.533) | -6.68 (36.687) | -17.24 (35.159) | -14.30 (42.346) | -12.84 (44.818)
  Week 8: number analyzed (Participants) | 67 | 66 | 67 | 71 | 35 | 62
  Week 8 | -20.37 (38.202) | -19.07 (39.531) | -12.99 (54.065) | -20.40 (36.544) | -25.58 (44.885) | -17.22 (41.533)
  Week 12: number analyzed (Participants) | 67 | 66 | 63 | 70 | 36 | 58
  Week 12 | -27.85 (44.630) | -19.14 (47.984) | -5.42 (61.699) | -23.68 (37.052) | -18.28 (69.762) | -20.35 (46.029)
  Week 16: number analyzed (Participants) | 66 | 65 | 64 | 68 | 37 | 63
  Week 16 | -34.70 (41.593) | -13.27 (54.785) | -19.75 (46.292) | -20.97 (42.685) | -25.05 (64.982) | -21.56 (47.588)

31. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥4 in the POEM Score, of Those With a Score of ≥4 at Baseline
Description: The efficacy of EDP1815 will be measured by the number of participants achieving a reduction of ≥4 in the POEM score, of those with a score of ≥4 at baseline at Week 16. There are 7 questions scored from 0 (no days) to 4 (every day), giving a POEM score range from 0 to 28, with higher scores representing higher disease severity.
Time Frame: 16 weeks
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 - Active: Participants with mild, moderate or severe Atopic Dermatitis who received placebo oral capsules. Participants with mild, moderate or severe Atopic Dermatitis who received 2 capsules (1.6 x 10^11 total cells) of EDP1815 (an orally administered, pharmaceutical preparation of a single strain of bacteria) once daily for 16 weeks.
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 66 | 66 | 65 | 72 | 37 | 66
Participants | 41 | 24 | 26 | 26 | 20 | 27

32. Secondary Outcome: Number of Courses of Rescue Therapy Per Participant
Description: The efficacy of EDP1815 will be measured by the number of rescue therapy courses per participant at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: Participants who received rescue therapy at each study visit listed were included as part of the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 75 | 74 | 74 | 86 | 38 | 74
Participants
  Week 4: number analyzed (Participants) | 75 | 72 | 74 | 81 | 38 | 74
  Week 4: 0 | 61 | 58 | 59 | 58 | 25 | 58
  Week 4: 1 | 5 | 6 | 5 | 12 | 6 | 4
  Week 4: 2 | 6 | 5 | 6 | 7 | 1 | 6
  Week 4: 3 or more | 3 | 3 | 4 | 4 | 6 | 6
  Week 8: number analyzed (Participants) | 68 | 66 | 66 | 72 | 38 | 66
  Week 8: 0 | 55 | 59 | 52 | 59 | 32 | 50
  Week 8: 1 | 6 | 4 | 8 | 5 | 2 | 3
  Week 8: 2 | 6 | 2 | 5 | 4 | 1 | 9
  Week 8: 3 or more | 1 | 1 | 1 | 4 | 3 | 4
  Week 12: number analyzed (Participants) | 64 | 62 | 59 | 68 | 37 | 64
  Week 12: 0 | 59 | 55 | 47 | 54 | 29 | 55
  Week 12: 1 | 3 | 3 | 6 | 6 | 4 | 4
  Week 12: 2 | 2 | 4 | 6 | 4 | 2 | 1
  Week 12: 3 or more | 0 | 0 | 0 | 4 | 2 | 4
  Week 16: number analyzed (Participants) | 63 | 55 | 54 | 64 | 36 | 58
  Week 16: 0 | 62 | 53 | 51 | 58 | 35 | 53
  Week 16: 1 | 1 | 2 | 3 | 3 | 0 | 3
  Week 16: 2 | 0 | 0 | 0 | 2 | 0 | 1
  Week 16: 3 or more | 0 | 0 | 0 | 1 | 1 | 1

33. Secondary Outcome: Number of Days of Treatment With Rescue Therapy Per Participant
Description: The efficacy of EDP1815 will be measured by the number of rescue therapy treatment days per participant at Weeks 1-8 and 9-16
Time Frame: 16 weeks
Population: All participants who received rescue therapy during the study were included as part of the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 75 | 74 | 74 | 86 | 38 | 74
Participants
  Weeks 1-8: number analyzed (Participants) | 75 | 72 | 74 | 81 | 38 | 74
  Weeks 1-8: 0 | 54 | 55 | 53 | 55 | 25 | 54
  Weeks 1-8: 1-7 | 10 | 8 | 9 | 16 | 5 | 8
  Weeks 1-8: 8-14 | 9 | 7 | 7 | 4 | 5 | 8
  Weeks 1-8: 15-21 | 2 | 2 | 2 | 4 | 1 | 1
  Weeks 1-8: 22 or more | 0 | 0 | 3 | 2 | 2 | 3
  Week 9-16: number analyzed (Participants) | 64 | 62 | 59 | 68 | 37 | 64
  Week 9-16: 0 | 53 | 51 | 42 | 50 | 27 | 48
  Week 9-16: 1-7 | 8 | 7 | 8 | 7 | 5 | 6
  Week 9-16: 8-14 | 2 | 4 | 9 | 8 | 4 | 7
  Week 9-16: 15-21 | 1 | 0 | 0 | 2 | 1 | 1
  Week 9-16: 22 or more | 0 | 0 | 0 | 1 | 0 | 2

34. Secondary Outcome: Proportion of Participants Not Requiring Rescue Therapy
Description: The efficacy of EDP1815 will be measured by the proportion of participants not requiring rescue therapy at Weeks 4, 8, 12 and 16
Time Frame: 4, 8, 12, and 16 weeks
Population: Participants who did not receive rescue therapy at any of the study visits were included as part of the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3 - Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Placebo | Cohort 4 - Active
Number analyzed (Participants) | 75 | 74 | 74 | 86 | 38 | 74
Participants
  Week 4: number analyzed (Participants) | 75 | 72 | 74 | 81 | 38 | 74
  Week 4 | 61 | 58 | 59 | 58 | 25 | 58
  Week 8: number analyzed (Participants) | 68 | 66 | 66 | 72 | 38 | 66
  Week 8 | 55 | 59 | 52 | 59 | 32 | 50
  Week 12: number analyzed (Participants) | 64 | 62 | 59 | 68 | 37 | 64
  Week 12 | 59 | 55 | 47 | 54 | 29 | 55
  Week 16: number analyzed (Participants) | 63 | 55 | 54 | 64 | 36 | 58
  Week 16 | 62 | 53 | 51 | 58 | 35 | 53

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected after the participant signing of the informed consent form (ICF) through 16 weeks of treatment plus an additional 28 days after taking their last dose of study drug.
Groups:
- All Placebo: Placebo participants from all cohorts
- Cohort 1 - Active: Mild, moderate or severe Atopic Dermatitis participants receiving 2 capsules (1.6 x 10^11 total cells) of EDP1815 once daily for 16 weeks.
Arm/Group | All Placebo | Cohort 1 - Active | Cohort 2 - Active | Cohort 3 - Active | Cohort 4 - Active
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/74 | 0/74 | 0/85 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/113 | 2/74 | 2/74 | 1/85 | 0/74
Other Adverse Events (participants affected / at risk) | 36/113 | 21/74 | 25/74 | 31/85 | 18/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Placebo (N=113) | Cohort 1 - Active (N=74) | Cohort 2 - Active (N=74) | Cohort 3 - Active (N=85) | Cohort 4 - Active (N=74)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis Toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Placebo (N=113) | Cohort 1 - Active (N=74) | Cohort 2 - Active (N=74) | Cohort 3 - Active (N=85) | Cohort 4 - Active (N=74)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5) | 5 (5) | 4 (4) | 2 (3)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4) | 4 (4) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 9 (9) | 7 (11) | 2 (2) | 3 (4) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (4) | 5 (5) | 2 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 (16) | 7 (7) | 14 (17) | 14 (17) | 4 (5)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (3) | 1 (1) | 3 (3) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the study, the data may be considered for reporting at a scientific meeting or for publication in a scientific journal. The sponsor has final approval authority over publication of the study data.

DOCUMENTS (2):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT05121480/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT05121480/SAP_001.pdf